CLINICAL TRIAL: NCT02876120
Title: The STavanger osteoARThritis Study in Primary Health Care
Brief Title: The STavanger osteoARThritis Study
Acronym: START
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diakonhjemmet Hospital (Other)
Collaborators: Stavanger Municipality (Unknown); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Nina Osteras, Senior researcher, Diakonhjemmet Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2016/1335
Record Dates: First submitted 2016-08-15; First posted 2016-08-23 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pre- and post-implementation phases (Other): Pre-implementation phase: during the pre-implementation period persons with hip or knee osteoarthritis will receive "usual care" as it is currently delivered by physiotherapists and general practitioners.
  Post-implementation phase: during the post-implementation phase the GPs and PTs will treat persons with hip or knee osteoarthritis according to the START treatment model including providing information/patient education program, supervised exercise and advice/support to loose weight and other non-surgical evidence based treatments modalities prior to being referred to an orthopaedic surgeon
  Interventions: Other: Implementation

INTERVENTIONS:
Other: Implementation — Multifaceted implementation strategy to implement evidence based international osteoarthritis treatment recommendations among GPs and PTs in private practice, template for PT discharge reports to GP, patient osteoarthritis education programs, and facilitate multidisciplinary collaboration between the PTs and GPs.

SUMMARY:
The START study will implement osteoarthritis (OA) treatment recommendations to increase the use of recommended treatment modalities and reduce non-desired events (e.g. unnecessary referrals to secondary care, unnecessary use of costly imaging modalities and use of treatment modalities supported by low quality of evidence). The purpose of the STavanger osteoARThritis (START) study is to improve the quality of OA care and increase the collaboration between health care professionals in primary health care and across health care levels.

DETAILED DESCRIPTION:
Previous research has shown that the osteoarthritis care for persons with hip or knee osteoarthritis in Norway has a potential for improvement as the provided care may not necessarily reflect evidence-based guideline recommendations. The purpose of the STavanger osteoARThritis (START) study is to improve the quality of OA care and increase the collaboration between health care professionals in primary health care and across health care levels.

Based on international treatment recommendations for OA care and previous research, a tailored implementation strategy targeting high quality, integrated care for people with OA in Stavanger Municipality will be developed, implemented and evaluated. The care will mainly be provided in the Stavanger primary health care services by physiotherapists (PT) (in private practice) and general practitioners (GP), but will also include collaboration with orthopaedic surgeons in specialist health care at Stavanger University Hospital.

The main aim of the present study is to develop, implement and evaluate effects of a tailored implementation strategy for the START study in Stavanger Municipality.

To evaluate the effects of the START implementation strategy, an interrupted time series design method will be applied. The study period will be divided into three phases: pre-implementation, implementation/transition and post-implementation. Data will be collected at 16 time points; 8 before and 8 after the implementation/ transition phase.

ELIGIBILITY:
Inclusion Criteria:

* PT working in private practice in Stavanger Municipality
* GP working in Stavanger Municipality
* Person with complaints due to hip and/or knee osteoarthritis referred to physiotherapy in Stavanger Municipality
* Person with complaints due to hip and/or knee osteoarthritis referred for assessment of joint replacement at Stavanger University Hospital

Exclusion Criteria:

* Persons referred to physiotherapy after a total joint replacement
* Persons who do not understand the Norwegian language
* Persons with cognitive dysfunction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported quality of osteoarthritis care | 8 weeks pre-implementation vs. 8 weeks post-implementation
  Using the "OsteoArthritis Quality Indicator questionnaire"

SECONDARY OUTCOMES:
Change in the number of PT discharge summaries to the referring GP | 8 weeks pre-implementation vs. 8 weeks post-implementation
Change in the proportion of people with OA referred to orthopaedic surgeon in secondary care that has explored non-surgical treatment modalities beforehand | 8 weeks pre-implementation vs. 8 weeks post-implementation
Change in the proportion of people with OA referred to orthopaedic surgeon in secondary care that has taken an MRI and/or conventional radiographs for OA assessment | 8 weeks pre-implementation vs. 8 weeks post-implementation
Change in the proportion of people with OA referred to orthopaedic surgeon in secondary care that leads to scheduled joint surgery | 8 weeks pre-implementation vs. 8 weeks post-implementation

CONTACTS AND LOCATIONS:
Overall Officials: Nina Østerås, Principal Investigator — Diakonhjemmet Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osteras N, Blaker IB, Hjortland T, Cottrell E, Quicke JG, Dziedzic KS, Blackburn S, Paulsen A. Improving osteoarthritis management in primary healthcare: results from a quasi-experimental study. BMC Musculoskelet Disord. 2021 Jan 14;22(1):79. doi: 10.1186/s12891-021-03959-6. PMID 33446167